CLINICAL TRIAL: NCT02447445
Title: Implementing Grip Strength Measurement Into Routine Clinical Practice; a Feasibility Study (GRImP)
Brief Title: Grip Strength Routine Implementation (GRImP)
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: RHM MED1250
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Frail Elderly, Inpatients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Older inpatient at MOP: The group includes older patients who are admitted to one of the Medicine for Older Patients (MOP) wards. Grip strength will be part of the routine assessment of older patient when admitted to MOP.
  Interventions: Procedure: Grip strength assessment

INTERVENTIONS:
Procedure: Grip strength assessment — Grip strength will be measured by the ward nurse using a Jamar dynamometer by asking the patient to squeeze with each hand twice, starting with the right hand using the standardised protocol The maximum GS measurement will be recorded. Patients who have low maximum GS values (men < 27 kg and women <16 kg) or those who are unable to perform the test will receive a care plan. The care plan will focus on review of dietary energy and protein intake and any need for oral nutritional supplements or dietetic review, and review of mobility with any need for physiotherapy review with regard to progressive resistance exercises to increase muscle strength.

SUMMARY:
Hand grip strength (GS) is a non-invasive marker of whole body skeletal muscle strength and function used in research and recommended as a simple inexpensive measure suitable for clinical use. Research has shown that low GS in hospital inpatients is associated with poor healthcare outcomes including increased postoperative complications, longer length of stay, increased functional limitations and disability. Measuring GS on admission to hospital has the potential to identify people at risk of poor healthcare outcomes allowing early intervention including focus on nutrition and mobility. Yet, GS measurement is not routinely used in clinical practice. The aim of this study is to evaluate the implementation of GS measurement into routine clinical practice in Medicine for Older People wards at UHS.

DETAILED DESCRIPTION:
This implementation research involves mixed methods combining qualitative and quantitative elements. The first preliminary part of the study will define the current baseline practice in the MOP wards in University Hospital Southampton (UHS) with regard to the identification of patients at high risk of poor healthcare outcomes, inpatients' nutritional care and management of their mobility. For this purpose, an ethnographic approach (involving interviews, focus groups, and audit of clinical records) will be followed. Understanding how the healthcare system works will enable justification and integration of GS measurement in the routine practice in an effective way. Participants and situations will be sampled on a purposive basis which means "cases/participants are sampled in a strategic way to best answer the research question". Single in-depth semi structured interviews will be conducted with different groups of healthcare staff with different levels of experiences and roles including consultants, junior doctors, ward sisters, dieticians, physiotherapists, and therapy assistants (a total of 10-15 healthcare staff members). The investigators will also conduct focus groups with nursing staff from the 5 wards, with nurses of similar seniority in each group to encourage free discussion (approximately 15-20 nurses divided into 4-5 focus groups) to gain an understanding of their shared practice.

The medical notes for the patients in the first 1-3 beds in each bay in the 5 wards will be examined (approximately 54 records). Basic information about the patient such as: age, gender, date of admission, domicile status, and reasons for admission will be first extracted. Then investigators will check the records to extract any information within the first 2-3 days of admission about risk assessment measures and what could indicate risk factors for poor healthcare outcomes. In addition, the number of and reasons for referrals weekly for the last 3 months to the dietetic team will be abstracted from the E-referral system. The number of prescribed oral nutritional supplements (ONS) will be also calculated weekly for the last 3 months from the electronic prescribing system. These figures are important for later analysis and comparison in order to assess changes in routine practice.

The second part of the research involves developing a training programme on measuring GS and creation of a care plan for older patients with low GS levels. Then, the nursing, medical and therapy staff in 5 wards in the MOP department will be trained in the measurement of grip strength and interpretation of grip strength values. There are approximately 150 nursing staff in MOP across the 5 wards, all of whom will be trained over a period of 3 months in GS measurement in groups of 5-10 each. Additional training sessions will be provided to junior doctors, consultants and therapy staff taking the opportunity to incorporate this into regular educational sessions where possible. The time and date of the training sessions will be defined and agreed liaising with the training lead in the MOP to avoid any disruption to the daily tasks of the MOP staff. The training session will last for approximately 1 hour. At the end of each session, participants will be asked to evaluate the training session using 5-points rating scale and give feedback. Nurses attending the training session will be asked as part of the training program to measure GS of a colleague according to the standard protocol as an assessment of their competency to measure GS of patients.

Implementation of GS should be start soon after completing the first training session in each ward. GS will be measured on all patients admitted to the MOP wards within 1-3 days of admission by a ward nurse. Only patients who are unable to squeeze the dynamometer handle such as patients with arthritis or who are very ill will be excluded. Grip strength will be measured by the ward nurse using a Jamar dynamometer by asking the patient to squeeze with each hand twice, starting with the right hand using the standardised protocol. A brief break of approximately 1 minute will be allowed between each squeeze. The maximum GS measurement will be recorded. A total of 5 Jamar dynamometers will be available for this study, one in each ward. The maximum GS values will be coded in two categories: score 1 representing values less than 27 kg for men and less than 16 kg for women which refers to patients at high risk of poor health outcomes, and score 2 representing values ≥27 kg for men and ≥16 kg for women representing lower risk. Patients who have low maximum GS values (men < 27 kg and women <16 kg) or those who are unable to perform the test will receive a care plan. The care plan will focus on review of dietary energy and protein intake and any need for oral nutritional supplements or dietetic review, and review of mobility with any need for physiotherapy review with regard to progressive resistance exercises to increase muscle strength.

During the implementation process, monitoring and evaluation of the outcomes of implementation which are referred to by the World Health Organisation (WHO) as "implementation outcome variables" will include assessing: acceptability of GS measurement, its adoption, coverage, fidelity, and costs.

Patients and staff acceptability will be assessed by conducting qualitative research (interviews or focus groups). A sample of 10-15 patients and 10-20 MOP staff is deemed to be enough to gain an understanding of their views and experience of GS measurement. Staff interviews will also assist understanding how GS routine implementation has been adopted and initiated in each of the five wards. Random weekly visits to MOP will be conducted to check fidelity and continuing staff competency on measuring GS as well as to audit the number of the number and proportion of patients who have their GS measured and those who have received a care plan in each ward. Coverage of GS implementation will be measured by calculating in the total number and proportion of patients who have their GS measured and those who have received a care plan in MOP within 6 months of routine implementation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be older patients admitted to the MOP.

Exclusion Criteria:

Exclusion criteria will be an inability to hold the dynamometer in either hand (eg pain and/or severe arthritis), inability to understand the explanation given (eg severe dementia or delirium), and terminal phase of illness.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Grip strength of older patients admitted to the MOP will be measured by a ward nurse.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The feasibility and acceptability of routine implementation of grip strength assessment in older patients | 6-9 months
  is it feasible to implement grip strength assessment routinely in Medicine for Older People (MOP) wards ? This will be determined by recording the proportion of older inpatients admitted to MOP wards who had their grip strength been measured and the percentage among them with low grip strength levels. The acceptability of routine implementation of grip strength will be assessed through qualitative method (interviews and focus groups) with older inpatients, medical staff, nursing staff, therapy and dietetic teams.

SECONDARY OUTCOMES:
The proportion of referrals to dietetic teams and the proportion of nutritional supplements prescriptions | After 3 months of routine implementation of grip strength
  When routine GS measurement has been implemented and embedded in clinical practice for at least 3 months, the number (or percentage) and reasons for referrals to the dietetic weekly for the preceding 3 months will be extracted from the E-referrals and will be compared to the numbers collected at the baseline. The number (or percentage) of ONS prescriptions will also be calculated from electronic prescribing system and compared to the baseline figures.
Costs of implementing grip strength assessment routinely in MOP | 9-12 months
  A cost analysis will include the implementation costs and NHS resource utilisation. The implementation costs will involve cost of equipment, recalibration, nurses training by band, and note audits. Resource use information will be collected as part of the study and those will include: nutritional prescriptions, referral to dietician, length of stay and discharge destination. The results will be presented as cost per patient detected and cost per unit of 120 beds.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Roberts, PhD, Study Chair — University General Southampton UHS
Locations (1):
- Southampton Genral Hospital, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ibrahim K, May CR, Patel HP, Baxter M, Sayer AA, Roberts HC. Implementation of grip strength measurement in medicine for older people wards as part of routine admission assessment: identifying facilitators and barriers using a theory-led intervention. BMC Geriatr. 2018 Mar 22;18(1):79. doi: 10.1186/s12877-018-0768-5. PMID 29566673
- See also: study protocol — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-016-0067-x
- See also: the study main findings — https://www.ncbi.nlm.nih.gov/pubmed/29566673